CLINICAL TRIAL: NCT06761027
Title: mFOLFIRINOX Combined With Anlotinib and Sintilimab as First-Line Therapy for Locally Advanced or Metastatic Pancreatic Cancer: A Prospective, Single-arm, Multicenter, Phase Ib/II Clinical Study
Brief Title: mFOLFIRINOX Plus Anlotinib and Sintilimab for Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Mao-Lin Yan, Department of Hepatobiliary Pancreatic Surgery, Fujian Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEC-SG-029-3.0
Record Dates: First submitted 2024-12-28; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: anlotinib; sintilimab
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mFOLFIRINOX Plus Anlotinib and Sintilimab (Experimental): Phase Ib: 6 patients will receive treatment at dose level-0 and their toxicity will be observed. If 2 or fewer patients experience dose-limiting toxicity, the study will proceed to the phase II part using dose level-0 as the treatment dose. If 3 or more patients have dose-limiting toxicity, another 6 patients will be accrued at a lower dose (dose -1). If two or fewer patients have dose-limiting toxicity, then we proceed with the phase II trial at that dose; otherwise, the trial is discontinued.
  Dose level - 0: anlotinib at a dose of 10mg per administration, once daily, orally administered on days 1-14, every 3 weeks.
  Dose level -1: anlotinib at a dose of 8mg per administration, once daily, orally administered on days 1-14, every 3 weeks.
  Phase II: The efficacy and safety of mFOLFIRINOX combined with anlotinib and sintilimab as first-line treatment for locally advanced or metastatic pancreatic cancer will be conducted at the anlotinib safe dose determined in phase Ib.
  Interventions: Drug: Anlotinib combined with Sintilimab

INTERVENTIONS:
Drug: Anlotinib combined with Sintilimab — Based on the mFOLFIRINOX chemotherapy regimen, combined with the safe dose of anlotinib determined in phase Ib and sintilimab.

SUMMARY:
This study is a prospective, single-arm, multicenter, phase Ib/II clinical trial that treats previously untreated patients with locally advanced or metastatic pancreatic cancer using mFOLFIRINOX in combination with anlotinib and sintilimab. The purpose of this trial is to evaluate the efficacy and safety of this treatment regimen and to preliminarily explore the correlation between biomarkers and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand this study and voluntarily sign the informed consent form;
2. Age between 18 and 75 years inclusive, with no gender restrictions;
3. Patients with locally advanced or metastatic pancreatic cancer diagnosed by histology or cytology;
4. No prior anti-cancer treatment;
5. Patients must have at least one measurable lesion (according to RECIST 1.1 criteria);
6. ECOG PS score of 0-1;
7. Expected survival of at least 3 months;
8. No severe organic diseases of the heart, lungs, brain, liver, kidneys, or other organs;
9. Women of childbearing age must agree to use contraceptive measures during the treatment period and for 6 months after the end of treatment; negative serum or urine pregnancy test within 7 days before study enrollment, and must be non-lactating, men must agree to use contraceptive measures during the study period and for 6 months after the study ends.

Exclusion Criteria:

1. Have already received or are currently receiving additional anti-tumor treatment measures such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, or traditional Chinese medicine treatment;
2. Known allergies to any of the drugs in the study;
3. Symptomatic brain metastases or metastases with symptom control time less than 2 months;
4. A large liver metastasis burden, occupying more than 70% of the liver volume;
5. Patients with obstructive jaundice whose bilirubin cannot be reduced to the expected level after adequate decompression;
6. Presence of any active autoimmune diseases or patients with autoimmune diseases expected to relapse (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes);
7. History of immunodeficiency; patients currently using immunosuppressants, systemic corticosteroid therapy, or any other form of immunosuppressive treatment;
8. Known genetic or acquired bleeding tendencies (such as coagulation disorders) or thrombosis, such as hemophiliacs; currently using or have recently (within 10 days before the start of the study treatment) used full-dose oral or injectable anticoagulants or thrombolytic drugs for therapeutic purposes (preventive use of low-dose aspirin, low molecular weight heparin is allowed);
9. Serious infections (CTC AE greater than grade 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; baseline chest imaging suggests active pulmonary inflammation, presence of symptoms and signs of infection within 2 weeks before the first use of the study drug, or requiring oral or intravenous antibiotic treatment (excluding the use of antibiotics for prevention);
10. History of other malignant tumors within the past 5 years or concurrently, except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, and papillary thyroid carcinoma;
11. Patients with mental illness; history of abuse of psychotropic drugs, alcoholism, and drug addiction;
12. Pregnant or lactating women;
13. Deemed by the investigator as unsuitable to participate in this trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | Four weeks after the initiation of medication until the day before surgery
  The Objective response rate (ORR) was defined as the complete response (CR) rate or the partial response (PR) rate according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall survival, OS | From date of enrollment until the date of death from any cause, assessed up to 60 months
  The Overall survival (OS) was defined as the time between receiving treatment and observing death or loss of follow-up for any reason.
Progression free survival, PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The Progression free survival (PFS) was defined as the time between the start of treatment and the progression of intrahepatic and/or extrahepatic tumors, or the occurrence of death or loss of follow-up for any reason.
Disease control rate, DCR | Four weeks after the initiation of medication until the day before surgery
  The Disease control rate (DCR) was defined as the complete response (CR) rate or the partial response (PR) rate or stable disease (SD) rate according to RECIST v1.1.
Toxicity Adverse events | From the initiation of medication, with recordings made whenever an adverse reaction occurs, assessed up to 60 months
  Grade 1-5 AEs according to NCI-CTCAE V5.0.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Zhangzhou Affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian